CLINICAL TRIAL: NCT06511336
Title: Evaluation of Alkaline Water Effect on Salivary Streptococcus Mutans in Children
Brief Title: Alkaline Water and Salivary Bacterial Count
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, Inas Karawia, Lecturer at Pediatric and Community Dentistry Department, Faculty of Dentistry, Pharos University in Alexandria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UREAC-04-3-222
Record Dates: First submitted 2024-07-09; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Dental Caries
Keywords: streptococcus mutans; chlorohexidine; Alkaline water
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- children using Alkaline water as mouthwash (FLO- bottled natural drinking water - made in Egypt) (Experimental): Children in this group will be asked to use alkaline water as mouthwash once daily for 3 weeks
  Interventions: Drug: Alkaline water (FLO water- Bottled drinking water- the Egyption Saudi Company for natural water- made in Egypt
- children using chlorohexidine mouthwash (Orovex- MARCO Pharmaceuticals- made in Egypt) (Active Comparator): Children in this group will be asked to use chlorohexidine as mouthwash once daily for 3 weeks
  Interventions: Drug: Alkaline water (FLO water- Bottled drinking water- the Egyption Saudi Company for natural water- made in Egypt
- children using tap water as mouthwash (Placebo Comparator): Children in this group will be asked to use tap water as mouthwash once daily for 3 weeks
  Interventions: Drug: Alkaline water (FLO water- Bottled drinking water- the Egyption Saudi Company for natural water- made in Egypt

INTERVENTIONS:
Drug: Alkaline water (FLO water- Bottled drinking water- the Egyption Saudi Company for natural water- made in Egypt — children will use Alkaline water as mouthwash daily for 3 weeks. each time they will use 10 ml of their mouthwash for 30 seconds
  Other Names: Alkaline water

SUMMARY:
This study will be aimed to examine the effect of alkaline water on salivary streptococcus mutans bacteria which is the main cause of dental caries and comparing its effect with chlorohexidine mouthwash on the children aged 10-12. tap water will be used as mouthwash for negative control group.

DETAILED DESCRIPTION:
Oral health has a major influence on one's general and oral health-related quality of life and well-being. Dental caries is characterized by demineralization of calcified tissues of the teeth due to several factors. Approximately, 60-65% of children in India are affected by dental caries. Several organisms are involved in the development of carious lesions. However, the literature strongly reports Streptococcus mutans (S. mutans) as the potential organism involved in the initiation of dental caries. This is because S. mutans can attach to the enamel surface, produce acid metabolites, provide glycogen reserves, and can synthesize extracellular polysaccharides.

Several antimicrobial agents with varying efficacy have been reported for the reduction of dental caries. Preventive programs such as the use of fluoride toothpaste, community water fluoridation, and mouth rinses, focusing primarily on the reduction of caries have also been carried out to reduce the prevalence of the disease. These substances inhibit the adhesion of bacteria, their colonization, and metabolic activity ultimately affecting their growth. Presently, bisbiguanide being the most efficacious chemotherapeutic agent against S. mutans has high bactericidal activity against both gram-positive and gram-negative bacteria. But it has a few side effects such as tooth discoloration, the altered sensation of taste, and erosion of oral mucosa. Also, due to the developing antimicrobial resistance to the currently available antibiotics and chemotherapeutics, the implementation of alternative treatment options for oral diseases that are safer, effective, and economical are needed.

Among various natural alternatives which have been studied, alkaline water has gained great interest in dentistry. alkaline water can be a safer and cheaper alternative to chemical adjuncts. The use of mouthwash is quite widespread by the public because the mouthwash is sold freely in stores, supermarkets, or supermarkets, the public only knows the effects of mouthwash to prevent bad breath alone, without knowing the side effects when using for a long time. Based on the problem, the researcher is interested to know whether the alkaline solution has a function like the function of mouthwash that can inhibit streptococcus mutans Materials and Methods this double-blinded randomized control clinical study will be carried out at Pedodontic clinics in Pharos University. A total of 30 schoolchildren will be selected by convenience sampling method. Inclusion criteria involved children between 10 and 12 years of age without any systemic disorder, or presence of gingivitis-calculus.

Exclusion criteria involved children who were already using mouthwashes, history of oral prophylaxis within 6 months, and had fixed or removable orthodontic appliances or removable prostheses. Written informed consent will be obtained from parents of all selected children. The children will be randomly divided into 3 groups by computer-generated random sequence: Group A - alkaline water group, Group B - 0.2% CHX mouthwash group, and Group C - Tap water group. The bottles will be coded along with the written instructions to use before dispensing to the children. The coding was will be done by a person who was not involved in the study; so that the double blinding design of the study was maintained. The children will be provided with 140 ml of their respective mouthwashes for home use every week. The children and examiner will be blind to allocation, i.e., the type of mouthwash. All the selected children were demonstrated a correct method of using mouthwash according to the group that they were assigned to. Children were instructed to use 10 ml of mouthwash as prescribed (i.e., take 10 ml of the mouth rinse in the measuring cap, rinse for 30 s, and spit out twice daily for 21 days), under the parent's supervision. A printed timetable for 3 weeks will be given to the parents, and they were asked to put a checkmark on the form after rinsing to check the compliance of the instructions given. The bacterial count will be evaluated at baseline, week 1, week 2, and week 3

Statistical analysis:

Data will be tabulated and analyzed using SPSS software version 25

ELIGIBILITY:
Inclusion Criteria:

* children aged 10-12 years

Exclusion Criteria:

* Children wearing orthodontic appliances.
* suffering from systemic diseases, and taking corticosteroids.
* taking antibiotics for at least one month

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-10 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Salivary streptococcus mutans count | 3 weeks
  the count of salivary coccus mutans bacteria which is the main cause of dental cariea

CONTACTS AND LOCATIONS:
Overall Officials: Inas M Karawia, Principal Investigator — Pharos University in Alexandria
Locations (1):
- Pharos University in Alexandria, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No